CLINICAL TRIAL: NCT03992313
Title: Community Versus Facility-based Services to Improve the Screening of Active HCV Infection in Cambodia: a Cluster Randomized Controlled Trial
Brief Title: Community Versus Facility-based Services to Improve the Screening of Active HCV Infection in Cambodia
Acronym: Cam-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University of Health Sciences, Phnom Penh, Cambodia (Unknown); Hopital Paul Brousse (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Fondation Mérieux (Other); University of Marseille (Other); SESSTIM UMR1252 (Aix-Marseille Univ, INSERM, IRD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ANRS 12384
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis C; Testing
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facility-based testing intervention (Experimental): * mass information on the possibility to be tested in health centers for HCV infection by CHWs ( information sheet and dedicated leaflet provided)
  * signed consent form collected at this step
  * HCV testing done in one of the referrals health centers, using the SD Bioline HCV RDT on a finger stick capillary whole blood.
  * In case of positive HCV RDT, immediate blood sample collection done in health center and sent to Provincial Hospital to perform HCV RNA using GenXpert viral load assay on plasma.
  * Results sent back to the health center and nurses in charge to give result to the participant and to refer to care in case of active infection
  Interventions: Other: Facility-based HCV rapid test; Other: Plasmatic HCV viral load
- Community-based testing intervention (Experimental): * dedicated training for CHWs to do the SD Bioline HCV RDT on a finger stick capillary whole blood directly in the household of participant.
  * Information provided by the CHW (information sheet and a dedicated Leaflet)
  * Signed consent form collected at this step.
  * onsite visits planned with the head of village in charge to inform the population about the study
  * In case of positive HCV RDT, 5 blood spots collected immediately on DBS and sent to Phnom Penh (Rodolphe Merieux laboratory) for HCV RNA extraction and amplification (Omunis)
  * Results sent back to the referral health center and nurses in charge to give result to the participant and to refer to care in case of active infection
  Interventions: Other: Community-based HCV rapid test; Other: DBS HCV viral load

INTERVENTIONS:
Other: Community-based HCV rapid test — HCV rapid tests will be done in the village
  Arms: Community-based testing intervention
Other: Facility-based HCV rapid test — HCV rapid tests will be done in the health center
  Arms: Facility-based testing intervention
Other: Plasmatic HCV viral load — HCV viral load will be done in provincial hospital on plasma using GenXpert
  Arms: Facility-based testing intervention
Other: DBS HCV viral load — HCV viral load will be done in Phnom Penh by DBS using Omunis kit
  Arms: Community-based testing intervention

SUMMARY:
Objectives Principal objective: to compare the effectiveness of a community-based intervention to a facility-based intervention to improve the combined-testing uptake (Antibody + RNA) of HCV infection among general population aged more than 40 years old in Cambodia Secondary objectives

* To compare the HCV antibody testing uptake between the 2 arms for the eligible population
* To compare the active case detection rate between the 2 arms for the eligible population
* To compare the linkage to care between the 2 arms for those with active infection
* To compare the cost-effectiveness of the two strategies
* To evaluate the treatment uptake
* To evaluate the effectiveness and safety of a 12-week dual-therapy of direct-acting antiviral (DAA) treatment

DETAILED DESCRIPTION:
Methodology: two-arms cluster-randomized controlled trial. Clusters are defined as a group of 50 households

Expected enrolment : 8000 patients in 160 clusters, 80 villages in each of the 2 provinces (Kompong Cham and Siem Reap)

Intervention

Arm 1: Facility-based testing intervention A team of community Health Workers (CHWs) will prepare a schedule to visit the selected villages and provide mass information on the possibility to be tested in health centers for HCV infection. Information will be provided using information sheet and a dedicated leaflet. If the participant agrees to participate, the signed consent form will be collected at this step. HCV testing will be done in one of the referrals health centers. HCV screening will be done using the SD Bioline HCV RDT on a finger stick capillary whole blood. Results will be available in 15 minutes. In case of positive HCV RDT, an immediate blood sample collection will be done in health center and sent to Provincial Hospital to perform HCV RNA using GenXpert viral load assay on plasma. Results will be sent back to the health center and nurses will be in charge to give result to the participant and to refer to care in case of active infection

Arm 2: Community-based testing intervention After a dedicated training, CHWs will do the SD Bioline HCV RDT on a finger stick capillary whole blood directly in the household of participant. Information will be provided by the CHW using information sheet and a dedicated leaflet. If the participant agrees to participate, the signed consent form will be collected at this step before any RDT collection. In case of structural or societal barriers for household testing, it will be possible to provide testing in a specific location in the village. The onsite visits will be planned with the head of village who will be in charge to inform the population about the study. In case of absence of participant during the first visit, a second visit will be scheduled. In absence of participant during the second visit, no additional visit will be planned. In case of positive HCV RDT, 5 blood spots will be collected immediately on DBS, dried at ambient temperature and put in an individual plastic bag with the ID number and sent to Phnom Penh (Rodolphe Merieux laboratory) for HCV RNA extraction and amplification (Omunis). Results will be sent back to the referral health center and nurses will be in charge to give result to the participant and to refer to care in case of active infection.

Treatment phase For positive HCV RNA, a consultation in the Provincial Hospital will be planned. The Baseline assessment will include questionnaires (risk behaviours and socio-economic status), clinical exam, blood sampling and liver ultrasound. Symptomatic cirrhotic patients will be referred to a National Hospital in Phnom Penh to a hepatology department. For the others patients, DAA treatment using sofosbuvir and daclatasvir combination for 12 weeks (Cambodian Essential Medicine List 2018) will be proposed, after checking the result of creatinine and the possible drug-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* All persons aged more than 40 years old
* Residing in the study area
* Informed consent obtained with oral information given and explained and the consent form signed by the participant and the nurse hired by the study at the latest the time of the RDT realization

Exclusion Criteria:

* Known positive HCV status with previous HCV treatment
* Severe disease present at inclusion involving life threatening
* Concurrent participation in any other clinical study without written agreement of the two study teams

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7692 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Combined-testing uptake | 12 months
  Combined-testing uptake defined as the number of persons tested for HCV RDT AND HCV RNA and aware of their status among the total number of persons eligible residing in the region where the intervention takes place

SECONDARY OUTCOMES:
HCV antibody testing uptake | 12 months
  HCV antibody testing uptake defined as the number of persons tested for HCV RDT and aware of their status among the total number of persons eligible residing in the region where the intervention takes place
Active case detection rate | 12 months
  defined as the number of persons with HCV active infection (positive HCV Ab and positive HCV RNA) and results given and explained among the total number of persons eligible residing in the region where the intervention takes place (measured and compared between the 2 arms)
Linkage to care | 12 months
  the number of persons with at least one consultation in the Provincial Hospital among the estimated total number of persons with active infection residing in the region where the intervention takes place (measured and compared between the 2 arms)

OTHER OUTCOMES:
Treatment uptake | 18 months
  the number of people initiating HCV treatment among the total number of persons with active infection linked to care (measured for the total population and not compared)
Liver-related morbidity and mortality | 18 months
  Proportion of patients with decompensated cirrhosis, HCC (measured for the total population and not compared)
Sustained virologic response 12 | 18 months
  Proportion of patients with sustained virologic response 12 weeks after discontinuation of treatment (SVR12) (measured for the total population and not compared)
Treatment failure | 18 months
  Proportion of patients with treatment failure defined as absence of SVR12 or missing HCV-RNA at 12 weeks post-treatment (PT12) due to treatment discontinuation for AEs or death (measured for the total population and not compared)

CONTACTS AND LOCATIONS:
Overall Officials: Vonthanak Saphonn, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Jean-Charles Duclos-Vallee, PhD, Principal Investigator — Paul Brousse hospital
Locations (2):
- Cambodia (2):
  - Chrey Vean Health Center, Kampong Cham, Kampong Cham
  - Han Chey Health Center, Kampong Cham, Kampong Cham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khuon D, Sagaon-Teyssier L, Neth S, Saint S, Meyer L, Mosnier E, Molino D, Phoeung CL, Chhay C, Heang K, Mam S, Duclos-Vallee JC, Segeral O, Saphonn V. Community-based versus facility-based services to improve hepatitis C screening in Cambodia: a cluster randomized controlled trial (ANRS 12384 Cam-C study). Lancet Reg Health West Pac. 2025 Oct 8;63:101703. doi: 10.1016/j.lanwpc.2025.101703. eCollection 2025 Oct. PMID 41127705
- [Derived] Mosnier E, Segeral O, Neth S, Sagaon-Teyssier L, Khuon D, Phoeung CL, Mam S, Chhay C, Heang K, Duclos-Vallee JC, Saphonn V. Community Versus Facility-Based Services to Improve the Screening of Active Hepatitis C Virus Infection in Cambodia: The ANRS 12384 CAM-C Cluster Randomized Controlled Trial-Protocol for a Mixed Methods Study. JMIR Res Protoc. 2024 Nov 20;13:e63376. doi: 10.2196/63376. PMID 39566053